CLINICAL TRIAL: NCT06129344
Title: Comparative Effects of Manual Lymphatic Drainage and Therapeutic Ultrasound on Breast Engorgement in Postpartum Women: A Feasibility Pilot Study
Brief Title: Lymphatic Drainage Versus Ultrasound for Postpartum Breast Engorgement: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was lower than the target 153 due to the pandemic, with only 35 participants. Four dropped out due to pandemic restrictions and health issues. The study will still proceed with analysis.
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202203042
Record Dates: First submitted 2022-06-06; First posted 2023-11-13 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-11

CONDITIONS: Breast Engorgement; Lactation Disorders
Keywords: breast engorgment; breast care; ultrasound therapy; breast feeding; manual lymphatic drainage; physical therapy modalities; postpartum
MeSH Terms: conditions — Lactation Disorders; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This study assesses the effectiveness of manual lymphatic drainage and therapeutic ultrasound on postpartum breast engorgement, pain, and hardness. It explores these interventions' impact on psychosocial support for breastfeeding mothers and medical attention. The goal is to identify the most effective treatment and examine its acceptability among postpartum women. The research will evaluate the processes of participant recruitment, randomization, and outcome assessment to ensure proper implementation and anticipate challenges. Additionally, it will consider whether these interventions should be included in Taiwan's National Health Insurance benefits, focusing on their cost-effectiveness and potential clinical benefits to enhance maternal care quality.
Who Masked: Participant
Masking Description: Typically, participants are unaware whether they are receiving experimental treatment or a control (e.g., standard care). The researchers and medical staff are aware of the treatment allocation.
  Due to medical ethics, if there is related breast pain and discomfort, the medical staff will still relieve the patient's breast pain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymphatic Drainage Group (Experimental): Manual Lymphatic Drainage Group: Performed by physiotherapists trained by Dr. Vodder School and licensed in Lymphatic Consolidation Detoxification Therapy (CDT). The patient's treatment posture is to lie down. First, start with the neck lymphatic drainage technique. After performing bilateral axillary lymph node activation and lymphatic valve contraction, the bilateral breast lymph fluid is drained to the bilateral lymph nodes. The time is about 20 minutes. Assist in removing milk from both breasts for 15 minutes each. Once a day for three consecutive days of treatment.
  Interventions: Other: Manual Lymphatic Drainage Group
- Ultrasound therapy group (Experimental): Ultrasound therapy group: performed by a physical therapist. This study uses an ultrasonic therapy device (model: UTO US-750 Therapeutic Ultrasound), frequency: 1MHz, intensity set to 1.0 Watt/cm2, pulsed mode, duty cycle 100%, treatment time 2 5 minutes on each side, and then assist in removing the breast milk from both breasts for 15 minutes on each side. Once a day for three consecutive days of treatment.
  Interventions: Other: Ultrasound therapy group

INTERVENTIONS:
Other: Manual Lymphatic Drainage Group — Manual Lymphatic Drainage Group:Performed by physiotherapists trained by Dr. Vodder School and licensed in Lymphatic Consolidation Detoxification Therapy (CDT). The patient's treatment posture is to lie down. First, start with the neck lymphatic drainage technique. After performing bilateral axillary lymph node activation and lymphatic valve contraction, the bilateral breast lymph fluid is drained to the bilateral lymph nodes. The time is about 20 minutes. Assist in removing milk from both breasts for 15 minutes each. Once a day for three consecutive days of treatment.
  Arms: Manual Lymphatic Drainage Group
Other: Ultrasound therapy group — Ultrasound therapy group: performed by a physical therapist. This study uses an ultrasonic therapy device (model: UTO US-750 Therapeutic Ultrasound), frequency: 1MHz, intensity set to 1.0 Watt/cm2, pulsed mode, duty cycle 100%, treatment time 2 5 minutes on each side, and then assist in removing the breast milk from both breasts for 15 minutes on each side. Once a day for three consecutive days of treatment.
  Arms: Ultrasound therapy group

SUMMARY:
In this article, women were randomly assigned to the manual lymphatic drainage group, therapeutic ultrasound group, and control group, and the breast pain, swelling hardness, and milk excretion before and after each treatment were measured.

DETAILED DESCRIPTION:
Breast engorgement as the swelling and distention of breast, which is one of the most common problems of postpartum of 3-8 days. At the same time, the congested blood vessels and tissue fluid will enter the surrounding tissues, resulting in the retention of tissue fluid and blood, resulting in interstitial fluid. In cases such as interstitial edema, the flow of milk is restricted.

There are many conservative treatments for relieving breast swelling. At present, there have been published studies on the application of ultrasound therapy and manual lymphatic drainage to breast problems during lactation. Previous studies have shown that manual lymphatic drainage and ultrasound therapy can significantly improve the pain, temperature, and firmness of breast engorgement. Manual lymphatic drainage and ultrasound therapy have been widely used in physical therapy, but there is little empirical evidence for manual lymphatic drainage on breast swelling. It is hoped that this empirical medical research method can be used to reduce the effect of breast pain caused by breast problems and improve breast milk. The purpose of this study was to examine whether manual lymphatic drainage and ultrasound therapy can improve breast pain, breast swelling, and increase the flow and volume of milk removed.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* Physiological breast swelling, breast heaviness, lumps, milk plugging, breast pain after childbirth
* Able to read and understand Chinese
* At least four points on the Breast Swelling Scale

Exclusion Criteria:

* Autoimmune system problems
* physical and mental health problems
* Breast abscesses, mastitis
* Breast implants
* Cardiac pacemakers
* Malignant tumors

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The Breast Enhancement Assessment Scale | Change from Baseline The Breast Enhancement Assessment Scale at 3day
  There are six grades of breast swelling: grade 1: tender, the breast does not change; grade 2: slight change; grade 3: the breast feels thick without tenderness; grade 4: the breast feels thick and begins to pressure Pain; Grade 5: Thick breasts with obvious tenderness; Grade 6: Very hard and very painful.
The Visual Analogue Scale for Pain；VASP | Change from Baseline The Visual Analogue Scale for Pain；VASP at 3day
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10. A higher score indicates greater pain intensity.
The Total Daily Milk Volume | Change from Baseline The Total Daily Milk Volume at 3day
  Total Daily Milk Volume was be recorded.

SECONDARY OUTCOMES:
Increase breastfeeding rates | 3day
  Continued breastfeeding was measured by the yes or no Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: ya-chun chang, Study Chair — Researchers
Locations (1):
- TMU-Joint Institutional Review Board, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided